CLINICAL TRIAL: NCT06340230
Title: A Phase II Study of SHR-A1811 Alone or in Combination With Adebrelimab as Neoadjuvant Treatment in HR Positive/HER2 Low Breast Cancer
Brief Title: SHR-A1811 Alone or in Combination With Adebrelimab as Neoadjuvant Treatment in HR Positive/HER2 Low Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Caigang Liu, Director of the Cancer Center, Shengjing Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-NEO-IIT-SHR-A1811-SHR1316
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: HR Positive/HER2 Low Breast Cancer
Keywords: SHR-A1811; Adebrelimab; Neoadjuvant; HR Positive/HER2 Low Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (PD-L1 Positive) SHR-A1811 Injection + Adebrelimab Injection (Experimental): SHR-A1811 Injection + Adebrelimab Injection Drug: SHR-A1811 Injection Drug: Adebrelimab Injection
  Interventions: Drug: SHR-A1811 Injection + Adebrelimab Injection
- Arm 2 (PD-L1 Negative) SHR-A1811 Injection + Adebrelimab Injection (Experimental): SHR-A1811 Injection + Adebrelimab Injection Drug: SHR-A1811 Injection Drug: Adebrelimab Injection
  Interventions: Drug: SHR-A1811 Injection + Adebrelimab Injection
- Arm 3 SHR-A1811 Injection (Experimental): SHR-A1811 Injection Drug: SHR-A1811 Injection
  Interventions: Drug: SHR-A1811 Injection

INTERVENTIONS:
Drug: SHR-A1811 Injection + Adebrelimab Injection — Drug: SHR-A1811 Injection Drug: Adebrelimab Injection
  Arms: Arm 1 (PD-L1 Positive) SHR-A1811 Injection + Adebrelimab Injection
Drug: SHR-A1811 Injection + Adebrelimab Injection — Drug: SHR-A1811 Injection Drug: Adebrelimab Injection
  Arms: Arm 2 (PD-L1 Negative) SHR-A1811 Injection + Adebrelimab Injection
Drug: SHR-A1811 Injection — Drug: SHR-A1811 Injection
  Arms: Arm 3 SHR-A1811 Injection

SUMMARY:
This is an open-label, phase II study evaluating the efficacy and safety of SHR-A1811 alone or in combination with Adebrelimab in Stage II-III HR Positive/HER2 Low Breast Cancer. Subjects will receive the neoadjuvant therapy of SHR-A1811 alone or in combination with Adebrelimab for six cycles, and then undergo surgery within 4 weeks after neoadjuvant therapy. Efficacy will be assessed every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥ 18 but ≤ 75 years
2. Histologically confirmed to be HR+/HER2-Low invasive breast cancer
3. Treatment-naive patients with stage II-III
4. Eastern Cooperative Oncology Group (ECOG) score is 0 or 1
5. Good level of organ function
6. Subjects must participate voluntarily, sign the informed consent form, have good compliance, and cooperate with follow-up visits

Exclusion Criteria:

1. Previously been treated with any anti-tumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.)
2. Received any other anti-tumor therapy at the same time
3. Bilateral breast cancer, inflammatory breast cancer or occult breast cancer
4. Stage IV breast cancer
5. Not confirmed by histopathology
6. With a history of any malignancies in the past 5 years, excluding cured cervical carcinoma in situ and melanoma skin cancer
7. Participated in other drug clinical trials within 4 weeks before enrollment
8. Known allergic history of the drug components of this protocol
9. History of immunodeficiency
10. Clinically significant cardiovascular diseases
11. Known or suspected interstitial lung disease
12. Active hepatitis and liver cirrhosis
13. Known hereditary or acquired bleeding thrombotic tendency
14. History of neurological or psychiatric disorders

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response (tpCR: ypT0-is/ypN0) | At the time of surgery

SECONDARY OUTCOMES:
Breast pathological complete response (bpCR：ypT0-is) | At the time of surgery
Residual cancer burden (RCB) | At the time of surgery
Best overall response rate (BORR) | During 18 weeks of the neoadjuvant treatment
Overall survival (OS) | 5 years
Disease-free survival (DFS) | 5 years
Event-free survival (EFS) | 5 years
Health-related quality of life (HRQOL) (EORTC QLQ-C30) | During 18 weeks of the neoadjuvant treatment
  The European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) Core 30 (EORTC QLQ-C30)
Health-related quality of life (HRQOL) | During 18 weeks of the neoadjuvant treatment
  The European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire Breast Cancer (EORTC QLQ- BR23) will be used to measure the HRQOL

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, MD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning, China